CLINICAL TRIAL: NCT01213212
Title: Preventing Renal Functional Abnormalities Predisposing to Chronic Kidney Disease in Abdominal Obesity: A Randomized, Parallel-Group, Pilot Study of Calorie REstriction in Subjects With Abdominal Obesity and Type 2 Diabetes at Increased Renal and Cardiovascular Risk
Brief Title: Preventing Renal Functional Abnormalities With Calorie Restriction in Subjects With Abdominal Obesity and Type 2 Diabetes at Increased Renal and Cardiovascular Risk
Acronym: CRESO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Collaborators: Istituto Superiore di Sanità (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CRESO
Record Dates: First submitted 2010-09-30; First posted 2010-10-01 (Estimated); Last update posted 2013-02-21 (Estimated); Status verified 2013-02

CONDITIONS: Diabetes Mellitus
Keywords: Caloric restriction; type 2 diabetes; abdominal obesity; renal disease
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2; Obesity, Abdominal; Kidney Diseases | interventions — Caloric Restriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Caloric restriction (Experimental): Caloric restriction
  Interventions: Other: Caloric restriction
- Diet "ad libitum" (Sham Comparator): Diet "ad libitum"
  Interventions: Other: No intervention

INTERVENTIONS:
Other: Caloric restriction — Caloric restriction.
  Arms: Caloric restriction
Other: No intervention — Diet "ad libitum"
  Arms: Diet "ad libitum"

SUMMARY:
The study investigates whether a caloric restricted dietary regime can prevent onset and/or progression of chronic kidney disease in type 2 diabetic patients with abdominal obesity, through the amelioration of concomitant metabolic abnormalities such as insulin resistance, dyslipidemia, hypertension and inflammation, possible risk factors for the onset of kidney disease.

The main aim of the study is therefore to evaluate the renoprotective effect of caloric restriction (CR) on subjects at risk of nephropathy. Secondary aim is to better understand how dietary implementation can modulate renal disease and its associated metabolic abnormalities.

DETAILED DESCRIPTION:
Background:

Obesity is the major risk factor for type 2 diabetes, which in turn is associated with nephropathy in about one third of patients. Obesity is also an independent risk factor for chronic renal disease, regardless of the association with diabetes. Furthermore, chronic renal disease is the strongest risk factor for cardiovascular morbidity and mortality in people with diabetes and without. However, the mechanisms responsible for the adverse nephrologic effects of obesity and type 2 diabetes are not clear, but likely involve insulin resistance, low-grade systemic inflammation, hyperlipidemia, and increased synthesis of vasoactive and fibrogenic substances, including angiotensin II, insulin, leptin and transforming growth factor β1. These substances may individually or interactively affect glomerular hyperfiltration, renal venous pressure, mesangial cell hypertrophy and matrix production, ultimately leading to renal scarring, impaired glomerular filtration rate, micro- and macro- albuminuria and end-stage renal disease (ESDR). Of interest, the risk for glomerular hyperfiltration and hyperperfusion is enhanced especially in subjects with abdominal obesity. Both conditions predispose to microalbuminuria, an early marker of renal disease and increased cardiovascular risk.

A growing body of evidence is now showing that calorie restriction (CR) improves many of the metabolic abnormalities associated with obesity and type 2 diabetes. In particular, it was recently demonstrated that long-term CR results in profound and sustained beneficial effects on the major atherosclerosis risk factors, serum Total cholesterol, Low density lipoprotein (LDL)-C, High density lipoprotein (HDL)-C, triglycerides, and blood pressure. CR also provides a powerful protective effect against obesity, insulin resistance, inflammation, as reflected in extremely low C reactive protein (CRP) levels and tumor necrosis factor (TNF)-alpha, and cardiovascular aging itself (i.e. left ventricular stiffness). We also found that long-term CR reduces serum concentrations of proinflammatory cytokines, triiodothyronine and growth factors such as platelet-derived growth factor (PDGF), and transforming growth factor (TGF)-beta-1, also factors actively involved in the progression of chronic kidney diseases. Taken together, these preliminary evidences suggest that CR might prevent renal function deterioration in diabetic, obese patients. However, this hypothesis has not been tested so far.

Objectives:

* The major goal of this pilot, explorative study is to provide a comprehensive evaluation of the effects of CR on the pathophysiological mechanisms that may affect the onset and the progression of chronic kidney disease in subjects with abdominal obesity and type 2 diabetes.
* Evaluate whether CR reduces the glomerular filtration rate (GFR) in subjects with abdominal obesity and type 2 diabetes, but still no evidence of renal disease [serum creatinine <1.2 mg/dL and albuminuria <20 μg/min (median of the 3 consecutive measurements in overnight urine collections)], and to assess whether CR reduces also kidney perfusion and/or filtration fraction, and whether these hemodynamic changes correlate with a concomitant reduction in urinary albumin excretion rate.
* Investigate the relationships between the changes in renal hemodynamics and/or albuminuria and the concomitant changes in abdominal circumference, body weight, body mass index, blood pressure, insulin sensitivity (as assessed by euglycemic-hyperinsulinemic clamp), serum lipids, adipokines levels (namely adiponectin, leptin), angiotensin II, and markers of chronic inflammation.
* Assess whether CR may reduce risk factors for cardiovascular disease (CVD) in diabetic, obese patients (insulin resistance, visceral obesity, hypertension).

Design:

After a baseline evaluation of clinical (blood pressure, body weight, abdominal circumference) and routine laboratory parameters, renal hemodynamics [glomerular filtration rate (GFR) and renal plasma flow (RPF) assessed by iohexol and PAH plasma clearances, respectively, and filtration fraction (FF) and renal vascular resistance (RVR) calculated by standard formulas], insulin sensitivity (estimated by euglycemic-hyperinsulinemic clamp), full lipid profile assessments, and urinary albumin excretion rate (mean of three measurements in three consecutive overnight urine collections), patients satisfying the selection criteria will be randomly allocated to either the CR intervention (25% CR) or an "ad libitum" diet (AL) for 6 months. The dietary guidelines for the calorie restricted diet will be based on the measurement of the individual food-intake diary and "resting metabolic rate" (RMR) (measured using indirect calorimetry) at baseline. CR will correspond to a calorie decrease by 25% as calculated from the baseline calorie intake measured with a 7-days food-intake diary and "RMR x activity levels" (activity levels will be calculated using the physical activity questionnaire). A food-intake diary will be provided with specific instruction by the Investigator (in written form). Baseline evaluations will be repeated every three months until the end of the study (except the renal hemodynamics studies and the euglycemic-hyperinsulinemic clamp that will be repeated only at month 6).

ELIGIBILITY:
Inclusion Criteria:

* Age >40 years
* Type 2 diabetes (ADA criteria)
* Waist circumference > 94 cm (males) or > 80 cm (females)
* UAE <20 μg/min
* Serum creatinine < 1.2 mg/dL
* No major changes in calorie, protein and sodium intake and in concomitant treatments with blood pressure, glucose or lipid lowering agents
* Patients legally able to give written informed consent to the trial (signed and dated by the patient)
* Written informed consent.

Exclusion Criteria:

1. Concomitant non-diabetic renal disease:

   * ischemic kidney disease
   * primary or immune-mediated renal disease
   * urinary tract obstruction or infection.
2. Concomitant treatments or clinical conditions that may affects renal hemodynamics and/or albuminuria:

   * ACE inhibitors and/or angiotensin II receptor blockers /ARBs
   * steroids and/or non-steroid antiinflammatory agents
   * thiazide or loop diuretics that, on the basis of the Investigator's judgment, might sustain hypovolemia and/or sodium depletion (with secondary kidney hypoperfusion/hypofiltration)
   * heart failure and/or hemodynamically significant left ventricular systolic dysfunction, cirrhosis, uncontrolled hyperglycemia resulting in glycosuria, hyper/hypo natremia of any cause)
3. Other general conditions:

   * previous surgical procedures for weight loss
   * previous episodes of depression, or suicide attempts
   * chronic abuse of alcohol and drugs
   * pregnancy, ineffective contraception or peri-menopausal age
   * cancer or any chronic disease that might affect the completion of the study
   * any primary endocrinological diseases
   * unwillingness or inability to adhere to the rigors of the CR intervention over the entire 6-months intervention period
   * legal incapacity and/or other circumstances rendering the patient unable to understand the nature, scope and possible consequence of the trial
   * evidence of an uncooperative attitude
   * any evidence that patient will not be able to complete the trial follow-up
   * inability to fully understand the potential risks and benefit of the study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2009-09; Primary Completion 2012-12 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Glomerular Filtration Rate (GFR), absolute and percent change, at 6 months vs baseline. | 0 and 6 month.

SECONDARY OUTCOMES:
Renal Plasma Flow (RPF) | At baseline, 3 and 6 month
Filtration Fraction (FF) | At baseline, 3 and 6 month
Renal Vascular Resistance (RVR) | At baseline, 3 and 6 month.
Albuminuria | At baseline, 3 and 6 month.
Metabolic and inflammatory parameters. | At baseline and 6 month

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Center for Rare Diseases, Ranica, Bergamo, Italy